CLINICAL TRIAL: NCT05462496
Title: Pilot Study of Gut Microbiome Modulation to Enable Efficacy of Neoadjuvant Checkpoint-based Immunotherapy Following Chemotherapy in Pancreatic Adenocarcinoma
Brief Title: Modulation of the Gut Microbiome With Pembrolizumab Following Chemotherapy in Resectable Pancreatic Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Deirdre Cohen, Director, Gastrointestinal (GI) Oncology Program, Associate Professor of Medicine (Hematology and Medical Oncology),, Icahn School of Medicine at Mount Sinai
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY-21-01814
Record Dates: First submitted 2022-07-11; First posted 2022-07-18 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Pancreatic Cancer
Keywords: Pancreatic cancer; antibiotics; resectable; microbiome; pembrolizumab; chemotherapy
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Biopsy; folfirinox; Drug Therapy; Ciprofloxacin; Anti-Bacterial Agents; Metronidazole; pembrolizumab; Immunotherapy; Antibodies, Monoclonal; Pancreaticoduodenectomy; Pancreatectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Participants who had Chemotherapy Following Pancreatic Adenocarcinoma (Experimental): Participants to be given antibiotics and pembrolizumab, following chemotherapy for the treatment of surgically resectable pancreatic cancer.
  Interventions: Procedure: Biopsy; Drug: FOLFIRINOX; Drug: Ciprofloxacin; Drug: Metronidazole; Drug: Pembrolizumab; Procedure: Surgical Resection

INTERVENTIONS:
Procedure: Biopsy — Pre-treatment tumor biopsy
Drug: FOLFIRINOX — Patients will receive FOLFIRINOX chemotherapy every 2 weeks for 5 cycles. One cycle of mFOLFIRINOX = 14 days.
  Cycles of mFOLFIRINOX are delivered as follows*:
  * Oxaliplatin: 85 mg/m2 IV over 2 hours on Day 1, followed by,
  * Irinotecan: 150 mg/m2 IV over 90 minutes on Day 1, followed by,
  * Leucovorin**: 400 mg/m2 IV over 2 hours on Day 1, followed by,
  * 5FU: 2400 mg/m2 IV over 46-48 hours on Days 1-3
  Other Names: Chemotherapy
Drug: Ciprofloxacin — Ciprofloxacin and metronidazole will be initiated 7 days following 5th dose of FOLFIRINOX. Subjects will self-administer ciprofloxacin 500mg PO BID on days 1-21. Participants will be instructed to take the antibiotics with food to minimize stomach upset and to administer at the same time each day. Treatment with antibiotics will continue for 21 days unless there is unacceptable toxicity or disease progression. Subjects will record date, time and number of tablets they take on provided drug diaries.
  Other Names: Antibiotic
Drug: Metronidazole — Ciprofloxacin and metronidazole will be initiated 7 days following 5th dose of FOLFIRINOX. Subjects will self-administer metronidazole 500mg PO every 8 hours on days 1-21. Participants will be instructed to take the antibiotics with food to minimize stomach upset and to administer at the same time each day. Treatment with antibiotics will continue for 21 days unless there is unacceptable toxicity or disease progression. Subjects will record date, time and number of tablets they take on provided drug diaries.
  Other Names: Antibiotic
Drug: Pembrolizumab — Pembrolizumab will be initiated 7 days post initiation of antibiotics. Subjects will receive a flat dose of pembrolizumab 200mg IV over 30 minutes.
  Other Names: Immunotherapy; Monoclonal antibody
Procedure: Surgical Resection — Following completion of 21 days of antibiotics, participant will undergo repeat imaging studies. If there is no progressive disease which renders participant surgically unresectable (based on NCCN guidelines 2.2021), subject will undergo definitive surgical resection.
  Other Names: pancreaticoduodenectomy; pancreatectomy

SUMMARY:
A multi-institutional, single arm pilot study of antibiotics and pembrolizumab, following chemotherapy for the treatment of surgically resectable pancreatic cancer.

DETAILED DESCRIPTION:
Phase: Pilot Study Objectives

Primary Objectives:

• To determine the change in immune activation in pancreatic tumor tissue following treatment with antibiotics, pembrolizumab.

Secondary Objectives:

* To establish the safety and feasibility of pre-operative antibiotics in combination with pembrolizumab following chemotherapy
* To describe the preliminary anti-tumor activity of pre-operative therapy with antibiotics, pembrolizumab, and chemotherapy in subjects with resectable pancreatic cancer

Exploratory Objectives:

* To determine immunophenotypic changes in the pancreatic tumor microenvironment following depletion of the microbiome using antibiotics and inhibition of PD-1 with pembrolizumab and to correlate these changes with tumor response as measured by histologic regression.
* To determine changes in systemic immunogenicity as measured in PBMCs harvested from blood following depletion of the microbiome using antibiotics and inhibition of PD-1 with pembrolizumab and to correlate these changes with tumor response as measured by histologic regression.
* To determine changes in the microbiome as measured in tumor and stool following treatment with chemotherapy, antibiotics, and pembrolizumab and to correlate these changes with tumor response as measured by histologic regression.
* To correlate changes in immune activation with changes in microbiome abundance and composition.

Methodology: Multi-center, open label, single arm pilot study Endpoint

Primary endpoint:

• Achievement of immune response, defined as activation of one or more of the following T cell markers: HLA-DR, CD38, CD25, KI67, and CD69; activation is defined as an increase of 20% or more over baseline in percentage of T cells expressing the marker.

Secondary Endpoints:

* Adverse events graded according to the NCI's Common Terminology Criteria for Adverse Events (CTCAE v5.0).
* R0 resection rate and histologic regression score
* Histologic regression score
* Overall response rate (ORR)
* Overall survival rate (OS)

Exploratory Endpoints:

* Immune changes within blood and tissue following treatment and correlate with clinical endpoints
* Microbiome changes in tissue and stool following treatment and correlate with clinical and immunologic endpoints

Study Duration 5 years Participant Duration 6 months Enrollment Period 2 years Duration of IP administration 1 week

Study Centers/Sites Multicenter:

1. Mount Sinai Health System, Tisch Cancer Institute
2. TBD
3. TBD Number of participants: 25 participants with 11 accrued at Mount Sinai Health over 2 years Description of Study Agent/Procedure: Ciprofloxacin 500 mg PO BID days 63-84. Metronidazole 500 mg PO TID days 63-84. Pembrolizumab 200 mg IV day 70. 5-Fluorouracil 2400 mg/m2 IV 46-48 hours infusion days 1, 15, 28, 42, 56. Leucovorin 400 mg/m2IV days 1, 15, 28, 42, 56. Irinotecan 150 mg/m2IV days 1, 15, 28, 42, 56. Oxaliplatin 85mg/m2IV days 1, 15, 28, 42, 56. Key Procedures: Tumor biopsy, surgical resection, blood draws, and stool collection.

Statistical Analysis: The primary efficacy endpoint is the achievement of immune response, defined as activation of one or more of the following markers: HLA-DR, CD38, CD25, KI67, and CD69; activation is defined as an increase of 20% or more over baseline in percentage of cells expressing the marker. With 25 patients, a 95% exact confidence interval around the immune response rate will be no more than 0.46 units wide.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed pancreatic adenocarcinoma. Histologies other than adenocarcinoma, or any mixed histologies, will NOT be eligible. *Note: histology must be confirmed prior to study treatment, however, participants may be consented to study based on imaging results consistent with pancreatic adenocarcinoma and then undergo diagnostic and research biopsy simultaneously.
* Clinical stage T1-3, N0-2, M0 (per AJCC 8th ed)
* Resectable pancreatic cancer as defined by NCCN Guidelines 2.2021 and based on pancreatic protocol dual-phase CT imaging. Multi-detector computed tomography (MDCT) angiography, performed by acquiring thin, preferably sub-millimeter, axial sections using a dual-phase pancreatic protocol, with images obtained in the pancreatic and portal venous phase of contrast enhancement, is required.

  * No arterial tumor contact (celiac axis [CA], superior mesenteric artery [SMA], or common hepatic artery [CHA])
  * No tumor contact with the superior mesenteric vein (SMV) or portal vein (PV) or ≤180° contact without vein contour irregularity
* Age > 18 years
* Patients must agree to pre-treatment biopsy(which may have been collected on a universal consent), on-treatment biopsy, and definitive surgical resection
* ECOG performance status of 0 or 1
* No prior treatment for diagnosis of pancreatic cancer
* Normal organ and marrow function as defined below:

  * Absolute neutrophil count (ANC) ≥1500/µL
  * Platelets ≥100 000/µL
  * Hemoglobin ≥9.0 g/dL or ≥5.6 mmol/L (Criteria must be met without erythropoietin dependency and without packed red blood cell (pRBC) transfusion within last 2 weeks. )
  * Creatinine ≤1.5 × ULN OR Measured or calculated creatinine clearance (Creatinine clearance (CrCl) should be calculated per institutional standard., GFR can also be used in place of creatinine or CrCl) ≥30 mL/min for participant with creatinine levels >1.5 × institutional ULN; ; GFR=glomerular filtration rate; ULN=upper limit of normal .
  * Total bilirubin ≤1.5 ×ULN OR direct bilirubin ≤ULN for participants with total bilirubin levels >1.5 × ULN AST (SGOT) and ALT (SGPT) ≤2.5 × ULN; ALT (SGPT) =alanine aminotransferase (serum glutamic pyruvic transaminase); AST (SGOT) =aspartate aminotransferase (serum glutamic oxaloacetic transaminase);
  * International normalized ratio (INR) OR prothrombin time (PT) Activated partial thromboplastin time (aPTT) ≤1.5 × ULN unless participant is receiving anticoagulant therapy as long as PT or aPTT is within therapeutic range of intended use of anticoagulants

Note: This table includes eligibility-defining laboratory value requirements for treatment; laboratory value requirements should be adapted according to local regulations and guidelines for the administration of specific chemotherapies.

* Ability to understand and sign a written informed consent document. Participant must have willingness and ability to comply with scheduled visits, treatment plans, laboratory tests and other study procedures.
* A female participant is eligible to participate if she is not pregnant , not breastfeeding, and at least one of the following conditions applies:

  * Not a woman of childbearing potential (WOCBP) OR
  * A WOCBP who agrees to follow the study contraceptive guidance during the treatment period and for at least 120 days plus 30 days (a menstruation cycle) after the last dose of study treatment.
* Males who are sexually active with WOCBP must agree to follow study instructions for method(s) of contraception for the duration of treatment with study treatment(s) and for a total of 180 days post treatment completion. In addition, male participants must be willing to refrain from sperm donation during this time.

Exclusion Criteria:

* Borderline resectable, locally advanced or distant metastatic disease
* Any medical condition which makes definitive surgical resection of the pancreatic cancer contraindicated due to high risk of morbidity/mortality
* Has active autoimmune disease that has required systemic treatment in past 2 years (i.e., with use of disease-modifying agents, corticosteroids, or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment.
* Medical history and concurrent disease as below:

  -Participants with a condition requiring systemic treatment with either corticosteroids (> 10 mg
* Interstitial lung disease that is symptomatic or may interfere with the detection or management of suspected treatment-related pulmonary toxicity.
* Uncontrolled or significant cardiovascular disease including, but not limited to, any of the following:

  * Evidence of uncontrolled, active infection, requiring parenteral or oral anti-bacterial, anti-viral or anti-fungal therapy ≤ 28 days prior to screening on study.
  * Participants with a condition requiring chronic systemic oral treatment with either antibiotics or anti-fungals
  * Any uncontrolled inflammatory GI disease including Crohn's Disease and ulcerative colitis.
* Participants with active, known, or suspected autoimmune disease.
* Has received a live vaccine or live-attenuated vaccine within 30 days prior to the first dose of study drug. *Note: for those participants who will be undergoing planned splenectomy, vaccinations against S. pneumoniae, N. meningitidis, H. influenzae type b and influenza virus may be administered per standard practice.
* Use of probiotics ≤ 28 days prior to screening on study.
* Known human immunodeficiency virus (HIV), known active Hepatitis A, or known Hepatitis B
* History of acute diverticulitis within the last 6 months or current chronic diarrhea
* Expected to require any other form of antineoplastic or surgical therapy while on study.
* Pre-existing peripheral neuropathy > Grade 1, as defined by CTCAE v5.0.
* Pregnant or lactating women.
* A WOCBP who has a positive urine pregnancy test within 72 hours or no pregnancy test prior to registration.
* WOCBP who are unwilling or unable to use an acceptable method to minimize the risk of pregnancy for the entire study period and 120 days plus 30 days (a menstruation cycle) after the last dose of study treatment. WOCBP who are continuously not heterosexually active are also exempt from contraceptive requirements, but still must undergo pregnancy testing.
* Sexually active fertile men not using effective birth control if their partners are WOCBP.
* History of primary immunodeficiency.
* Has a history of (non-infectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease.
* History of organ allograft or allogeneic bone marrow transplant.
* Any prior radiation therapy, immunotherapy, or biologic ('targeted') therapy for treatment of the patient's pancreatic tumor. Biliary stent is allowed.
* Treatment for other invasive carcinomas within the last two years who are at greater than 5% risk of recurrence at time of eligibility screening. Carcinoma in-situ and basal cell carcinoma/ squamous cell carcinoma of the skin are allowed.
* Participation in any investigational drug study within 4 weeks preceding the start of study treatment.
* Major surgery, excluding laparoscopy, within 4 weeks of the start of study treatment, without complete recovery.
* History of allergy to study treatments or any of its components.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2023-03-16 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Achievement of overall immune response | at day 43
  Achievement of overall immune response, defined as activation of one or more of the following T cell markers: HLA-DR, CD38, CD25, KI67, and CD69; activation is defined as an increase of 20% or more over baseline in percentage of T cells expressing the marker. Comparison to be made between tissue biopsy taken following chemotherapy (and prior to antibiotics and pembrolizumab) and definitive surgical specimen.
Achievement of overall immune response | day 102
  Achievement of overall immune response, defined as activation of one or more of the following T cell markers: HLA-DR, CD38, CD25, KI67, and CD69; activation is defined as an increase of 20% or more over baseline in percentage of T cells expressing the marker. Comparison to be made between tissue biopsy taken following chemotherapy (and prior to antibiotics and pembrolizumab) and definitive surgical specimen.

SECONDARY OUTCOMES:
Adverse event incidence rate | at 6 months
  Adverse events will be graded according to the NCI's Common Terminology Criteria for Adverse Events (CTCAE v5.0)
R0 resection rate | at 3-4 months
  The R0 Resection Rate (percent) is defined as the percentage of resected specimen that have lateral and deep margins that are free of neoplasia under microscopic visualization.
Proportion of participants with histologic regression score 0, 1, or 2 | at 3-4 months
  The histologic regression score is defined as the proportion of patients with Grade 0, 1 or 2 histologic tumor response (Grade 0: no viable tumor; Grade 1: <5% viable tumor cells; Grade 2: ≥5% viable tumor cells)
Overall response rate (ORR) | at 3-4 months
  The overall response rate (ORR) is defined as the proportion of patients who achieve complete response (CR) or partial response (PR) as per the RECIST 1.1 criteria.
Overall survival rate (OS) | at 5 years
  Overall survival rate (OS) is defined as the duration of time from initial pembrolizumab administration to the date of death from any cause. Subjects who are alive or lost to follow-up as of the data analysis cutoff date will be censored for OS. The censoring date will be determined from the subject's date of last examination or data analysis cutoff date, whichever event occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: Deirdre Cohen, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: CSR
Time Frame: As soon as possible after publication - to be determined
Access Criteria: Researchers who provide a methodologically sound proposal. Any purpose. At Principal Investigator discretion (Deirdre.Cohen@mssm.edu)